CLINICAL TRIAL: NCT04915586
Title: Short Duration High Intensity Intrapleural Alteplase With Pulmozyme (DNase) in Pleural Infection Management- Single Centre Experience
Brief Title: Short Duration High Intensity Intrapleural Alteplase With Pulmozyme in Pleural Infection Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Mohamed Faisal Abdul Hamid, Associate Professor, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF-2020-008; NMRR-19-2940-51404 (Registry Identifier: Medical Research Ethic Committee of Ministry of Health Malaysia)
Record Dates: First submitted 2021-02-21; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Loculated Empyema
Keywords: Intrapleural fibrinolysis, pleural infection
MeSH Terms: interventions — dornase alfa; Deoxyribonucleases

STUDY DESIGN:
Masking Description: The radiologists were blinded to patient identity and intervention timing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Intra-pleural Alteplase 16mg with Pulmozyme (DNase) 5mg for total 3 doses within 24 hours
  Intervention Drug: Combination Alteplase and pulmozyme (DNase)
  Interventions: Drug: Intra-pleural Alteplase 16mg with Pulmozyme (DNase) 5mg

INTERVENTIONS:
Drug: Intra-pleural Alteplase 16mg with Pulmozyme (DNase) 5mg — Intra-pleural Alteplase 16mg with Pulmozyme (DNase) 5mg for total 3 doses within 24 hours
  Other Names: Combination Tissue Plasminogen Activator (t-PA) and Pulmozyme (DNase)

SUMMARY:
The aim of this study was to assess the efficacy of the modified regimen short duration intrapleural 16mg alteplase (Actilyse, Boehringer Ingelheim) with 5mg DNase (Pulmozyme Hoffmann-La Roche Ltd) in patients with pleural infection.

DETAILED DESCRIPTION:
The regimen 10 mg alteplase and 5 mg DNase twice daily that was used in MIST-2 trial is still an empiric choice. The rationale of using 3 doses of 16 mg alteplase dose (with supplementary 5 mg DNase) in our study was governed by the formulation of alteplase in our country (50 mg per ampoule); hence, it is best used within 24 hours following reconstitution as its biochemical stability up to 24 hours as assessed by in vitro clot lysis assays.

ELIGIBILITY:
Inclusion Criteria:

* adult patient with age more than 17 year old
* evidence of complex parapneumonic effusion or empyema; with poor pleural fluid drainage of ≤150 mL after 24 hours of insertion of chest drain
* clinical evidence of infection such as fever and or elevated C-reactive protein (CRP) or white-cell count
* complex pleural effusion proven by ultrasound
* pleural fluid analysis that fulfilled at least one of the characteristics: frank pus, exudative nature (according to light's criteria), gram stain or culture positive, lactate dehydrogenase (LDH) > 1000 U/L, pH < 7.2 and/or glucose level < 3.3mmol/L

Exclusion Criteria:

* known allergy to pulmozyme or alteplase
* acute stroke, active bleeding diathesis
* major surgery in past 5 days
* previous pneumonectomy on the infected side
* bronchopleural fistula
* pregnancy
* coagulopathy (INR > 2, APTT >100, platelet count < 50,000 cells)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Radiographic improvement in pleural opacity on chest radiograph | Day 7
  measured in percentage

SECONDARY OUTCOMES:
pleural fluid volume drained | Day 7
  measured in mls
changes in inflammatory markers C-Reactive Protein (CRP ) | Day 7
  reduction of inflammatory markers trend
White cell count | Day 7
  changes in inflammatory markers trend
length of hospitalisation | upto 30 days
  days
the need of surgical referral | upto 30 days
  if evidence of clinical deterioration post intrapleural therapy such as intrapleural haemorrhage or hypotension or less than 50% resolution of effusion on chest-xray post intrapleural therapy
adverse events post therapy | Day 7
  pain, bleeding events, hemodynamic stability
mortality rate at day 30 post intervention | 30 days
  days

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, Principal Investigator — Associate Professor
Locations (1):
- University Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Derived] Cheong XK, Ban AY, Ng BH, Nik Abeed NN, Nik Ismail NA, Nik Fuad NF, Syed Zakaria SZ, Ghan SL, Abdul Hamid MF. Modified regimen intrapleural alteplase with pulmozyme in pleural infection management: a tertiary teaching hospital experience. BMC Pulm Med. 2022 May 17;22(1):199. doi: 10.1186/s12890-022-01995-z. PMID 35581627